CLINICAL TRIAL: NCT02868593
Title: Etiology of Orphan Community-based Meningitis and Meningo-encephalitis.
Acronym: MENINGITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-47; 2013-A01538-37 (Other: ANSM)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Community-based Meningitis; Meningo-encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with clinical meningitis or meningo-encephalitis (Experimental)
  Interventions: Other: Pharyngeal swab

INTERVENTIONS:
Other: Pharyngeal swab

SUMMARY:
The primary purpose of this study is to assess the contribution of a non-invasive sampling (pharyngeal swab) in the diagnosis of community based meningitis or meningo-encephalitis.

DETAILED DESCRIPTION:
Community-based meningitis and meningo-encephalitis are defined by the presence of more than 10 leukocytes per mL of cerebrospinal fluid (CSF), eventually reported to the number of red blood cells. They can be associated with encephalitis, defined by cerebral or cerebellar dysfunction in the case of the transmission. The evolution includes death, what makes the seriousness of this clinical situation. However the diagnostic performance of meningitis and meningo-encephalitis in a patient without contact with a care structure is less than 25% resulting in empirical support in half of the patients. Indeed, the microbiological diagnosis of meningitis and transmission target currently only five pathogens including HIV positive resulted in a significant change to support the patient in three areas, decision of hospitalization, decision of isolation and antibiotic or antiviral treatment decision. A weekly epidemiological monitoring of the microbiological diagnosis of meningitis and meningo-encephalitis has enabled us to see a mismatch between a curve of requests for analyses and a flat curve of produced diagnoses. This discrepancy is interpreted as indicating a community outbreak of meningitis or meningo-encephalitis non-diagnosed by routine methods, called orphan meningitis or orphan meningo-encephalitis. On this observation, our research project is to improve the performance of the etiological diagnosis of community-based meningitis or meningo-encephalitis. To do this, we will evaluate the diagnostic performance of an advanced technique, using a non-invasive sample, the pharyngeal swab from the patient, to find micro-organisms that are not part of the commensal flora of the pharynx and who are responsible for undetected in routine meningitis. Indeed the main pathogens and meningitis (enterovirus, pneumococcus, meningococcus) transmission give a pharyngeal carriage before being responsible for meningitis or meningo-encephalitis. These bacteria are Coxiella burnetii, Bartonella spp., Tropheryma whipplei, Leptospira spp. and Borrelia spp.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged more than 18 years old.
* Patient with clinical meningitis or meningo-encephalitis with community transmission.
* Patient with a prescription of microbiological diagnosis of meningitis or meningo-encephalitis.
* Patient who do not declined to have his medical records reviewed for research
* Patient with health insurance

Exclusion Criteria:

* Minor Patient (age <18 years)
* Pregnant woman, parturient or breastfeeding
* Adult Patient under guardianship
* Patient deprived of liberty under court order
* Patient vital in emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with established etiological diagnosis of community based meningitis or meningo-encephalitis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided